CLINICAL TRIAL: NCT04608227
Title: Can Non-invasive Haemodynamic Monitoring With Clearsight(r) Predict Spinal Hypotension During Caesarian Section? A Prospective Observational Study
Brief Title: Non-invasive Haemodynamic Monitoring to Predict Spinal Hypotension During Caesarian Section
Status: Completed | Type: Observational
Sponsor: Hospital Nord (Other)
Responsible Party: Principal Investigator, Gary DUCLOS, Medical Doctor, Hospital Nord
Other Study IDs: Darnord-2020
Record Dates: First submitted 2020-10-19; First posted 2020-10-29 (Actual); Last update posted 2022-08-04 (Actual); Status verified 2022-08

CONDITIONS: Hypotension; Pregnancy Related; Spinal Anesthetics Causing Adverse Effects in Therapeutic Use
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Third trimester pregnant women undergoing ceasarean section
  Interventions: Device: Clearsight monitoring

INTERVENTIONS:
Device: Clearsight monitoring — Non invasive hemodynamic monitoring using a finger cuff Cardiac ultrasound performed to calculate Velocity - Time - integral (VTI) Both intervention are performed before and after a passive leg raising challenge.
  Other Names: Cardiac ultrasound

SUMMARY:
Spinal anaesthesia for elective caesarean section is associated with maternal hypotension, secondary to alteration of sympathetic tone and hypovolemia, in up to 70% of cases.

Our objective, in this prospective single-centre observational study, was to assess the ability of change in systolic ejection volume after 45° passive leg raising to predict hypotension after spinal anaesthesia. Systolic ejection volum was monitored with non-invasive Clearsight Device just before elective caesarean section in third trimester pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* third trimester pregnant women undergoing elective ceasarean section under spinal anesthesia

Exclusion Criteria:

* emergent ceasarean section
* eclampsia or pre-eclampsia
* undergoing anti-hypertensive treatment
* arythmia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only pregmant women
Study Population: prospective inclusion of 3 rd trimester pregnant women undergoing spinal anesthesia for elective ceasarean section
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-06-01 (Actual); Primary Completion 2020-11-26 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Systolic Ejection volume (mL) | 30 minutes
  Systolic ejection volume is measured using Clearsight (non invasive monitoring device)

SECONDARY OUTCOMES:
Velocity - Time - Integral (cm) | 30 minutes
  Velocity - Time - Integral is measured using transthoracic cardiac ultrasound

CONTACTS AND LOCATIONS:
Locations (1):
- Departement anesthesie reanimation hopital nord, Marseille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/35074676/